CLINICAL TRIAL: NCT02194790
Title: Effect of Integrated CKD Care Program in Early Diabetic Nephropathy in Primary Health Care Setting.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bhumirajanagarindra Kidney Institute, Thailand (Other)
Collaborators: Ministry of Health, Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CICC program
Record Dates: First submitted 2014-07-17; First posted 2014-07-18 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Chronic Kidney Disease; Diabetic Nephropathy
Keywords: Chronic Kidney Disease; Diabetic Nephropathy; Integrated Chronic Kidney Disease Care
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetic Nephropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- community-based Integrated CKD care (Experimental): Standard CKD care + multidisciplinary team and home visit by community care team
  Interventions: Behavioral: Community-based Integrated CKD Care
- Conventional CKD care (No Intervention): standard CKD care

INTERVENTIONS:
Behavioral: Community-based Integrated CKD Care — Patients received, in addition to the standard care, educational activities provided by nutritionist, pharmacist and physiotherapist, and quarterly home visits. Our home visits team consisted of nurse, health care officers and village health volunteers
  Other Names: Multidisciplnary clinic + home visit team
  Arms: community-based Integrated CKD care

SUMMARY:
Chronic kidney disease (CKD) is a major health problem in Thailand. Previous studies have demonstrated that integrated pre-dialysis care may slow the decline in renal function (Nephrol Dial Transplant.2009 Nov;24(11):3426-33). It is interesting to know whether early intervention especially in high risk groups like Diabetic may also improve outcome of these patients in primary health care setting resulting in delay of CKD progression.

DETAILED DESCRIPTION:
We conducted a 12-month longitudinal study at district A (control) and B (intervention) at Kamphaeng Phet Province, Thailand. Diabetic patients with eGFR ≥ 60 ml/min/1.73m2 were recruited from both districts. Patients in district A (control group) received standard CKD care according to NKF-K/DOQI guidelines1 whereas those in district B (intervention) received, in addition to the standard care, educational activities provided by nutritionist, pharmacist and physiotherapist, and quarterly home visits. Our home visits team consisted of nurse, health care officers and village health volunteers. During each hospital visit of both groups clinical data were assessed. All laboratory parameters were collected every 3 months, and LDL and HbA1C every 6 months. The primary end point was rate of eGFR decline. Secondary outcomes were random urine albumin to creatinine ratio (ACR), blood pressure, waist circumference, HbA1C and LDL .

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients with eGFR are equal or more than 60 ml/min/1.73m2 estimated twice at 3 months.

Exclusion Criteria:

* Active glomerular disease, obstructive uropathy, end-stage renal disease, HIV infection, pregnancy, body mass index (BMI) less than 18 or more than 40 kg/m2, being under treatment for malignancy, urine protein-creatinine ratio more than 3.5 g/g creatinine and active urinary sediment (urine red blood cells >3 cells/high power field or urine white blood cells >10 cells/high power field).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The difference of rate of estimated glomerular filtration(eGFR) decline | 12 months
  We compare the difference of rate of eGFR decline from baseline end of the study between the intervention group and control group.

SECONDARY OUTCOMES:
Change from baseline in Random Urine Albumin to Creatinine Ratio | 12 months
Change from baseline in waist circumference | 12 months
Change from baseline in low density lipoproteins(LDL) | 12 months
Change from baseline in systolic blood pressure | 12 months
Change from baseline in Hemoglobin A1C | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kotcharat Vipattawat, M.D., Principal Investigator — Bhumirajanagarindra Kidney Institute
Locations (1):
- Bhumirajanagarindra Kidney Institute, Bangkok, Bangkok, Thailand

REFERENCES:
- [Background] KDOQI. KDOQI Clinical Practice Guidelines and Clinical Practice Recommendations for Diabetes and Chronic Kidney Disease. Am J Kidney Dis. 2007 Feb;49(2 Suppl 2):S12-154. doi: 10.1053/j.ajkd.2006.12.005. No abstract available. PMID 17276798
- [Background] American Diabetes Association. Standards of medical care in diabetes--2012. Diabetes Care. 2012 Jan;35 Suppl 1(Suppl 1):S11-63. doi: 10.2337/dc12-s011. No abstract available. PMID 22187469
- [Background] Levin A, Stevens PE. Early detection of CKD: the benefits, limitations and effects on prognosis. Nat Rev Nephrol. 2011 Jun 28;7(8):446-57. doi: 10.1038/nrneph.2011.86. PMID 21712852
- [Background] Myers GL, Miller WG, Coresh J, Fleming J, Greenberg N, Greene T, Hostetter T, Levey AS, Panteghini M, Welch M, Eckfeldt JH; National Kidney Disease Education Program Laboratory Working Group. Recommendations for improving serum creatinine measurement: a report from the Laboratory Working Group of the National Kidney Disease Education Program. Clin Chem. 2006 Jan;52(1):5-18. doi: 10.1373/clinchem.2005.0525144. Epub 2005 Dec 6. PMID 16332993
- [Background] Black C, Sharma P, Scotland G, McCullough K, McGurn D, Robertson L, Fluck N, MacLeod A, McNamee P, Prescott G, Smith C. Early referral strategies for management of people with markers of renal disease: a systematic review of the evidence of clinical effectiveness, cost-effectiveness and economic analysis. Health Technol Assess. 2010 Apr;14(21):1-184. doi: 10.3310/hta14210. PMID 20441712
- [Background] Cueto-Manzano AM, Martinez-Ramirez HR, Cortes-Sanabria L. Comparison of primary health-care models in the management of chronic kidney disease. Kidney Int Suppl (2011). 2013 May;3(2):210-214. doi: 10.1038/kisup.2013.16. PMID 25018986
- [Background] Bayliss EA, Bhardwaja B, Ross C, Beck A, Lanese DM. Multidisciplinary team care may slow the rate of decline in renal function. Clin J Am Soc Nephrol. 2011 Apr;6(4):704-10. doi: 10.2215/CJN.06610810. Epub 2011 Jan 27. PMID 21273376
- [Background] Chobanian AV, Bakris GL, Black HR, Cushman WC, Green LA, Izzo JL Jr, Jones DW, Materson BJ, Oparil S, Wright JT Jr, Roccella EJ; National Heart, Lung, and Blood Institute Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure; National High Blood Pressure Education Program Coordinating Committee. The Seventh Report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure: the JNC 7 report. JAMA. 2003 May 21;289(19):2560-72. doi: 10.1001/jama.289.19.2560. Epub 2003 May 14. PMID 12748199
- [Result] Ingsathit A, Thakkinstian A, Chaiprasert A, Sangthawan P, Gojaseni P, Kiattisunthorn K, Ongaiyooth L, Vanavanan S, Sirivongs D, Thirakhupt P, Mittal B, Singh AK; Thai-SEEK Group. Prevalence and risk factors of chronic kidney disease in the Thai adult population: Thai SEEK study. Nephrol Dial Transplant. 2010 May;25(5):1567-75. doi: 10.1093/ndt/gfp669. Epub 2009 Dec 27. PMID 20037182
- [Result] Levey AS, Stevens LA, Schmid CH, Zhang YL, Castro AF 3rd, Feldman HI, Kusek JW, Eggers P, Van Lente F, Greene T, Coresh J; CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration). A new equation to estimate glomerular filtration rate. Ann Intern Med. 2009 May 5;150(9):604-12. doi: 10.7326/0003-4819-150-9-200905050-00006. PMID 19414839
- [Result] Kidney Disease Outcomes Quality Initiative (K/DOQI). K/DOQI clinical practice guidelines on hypertension and antihypertensive agents in chronic kidney disease. Am J Kidney Dis. 2004 May;43(5 Suppl 1):S1-290. No abstract available. PMID 15114537
- [Result] National Kidney Foundation. KDOQI Clinical Practice Guideline for Diabetes and CKD: 2012 Update. Am J Kidney Dis. 2012 Nov;60(5):850-86. doi: 10.1053/j.ajkd.2012.07.005. PMID 23067652